CLINICAL TRIAL: NCT00222144
Title: Phase II Study of Gleevec and Taxotere in Recurrent Non-Small Cell Lung Cancer
Brief Title: Study of Gleevec and Taxotere in Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Novartis (Industry); Kansas Masonic Cancer Research Institute (Unknown)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9698
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Imatinib Mesylate; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Gleevec and Taxotere
  Interventions: Drug: Gleevec and Taxotere

INTERVENTIONS:
Drug: Gleevec and Taxotere — Gleevec 600 mg QD for 12 months Taxotere IV 30 mg/m2 on day 1, 8 and 15
  Other Names: Docetaxel; Imatinib

SUMMARY:
The primary goal of this study is to determine the effects of the combination of Gleevec and Taxotere in lung cancer in terms of control and reduction of the cancer size. The study will also test lung cancer to see if the presence of certain protein called receptor for platelet derived growth factor can influence the effect of the treatment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the response rate of Gleevec with Taxotere in patients with recurrent non-small cell lung cancer. Also to determine the expression of PDGF-R, phosphorylated PDGF-r and C-kit in the original tissue and correlate with response. If the patient has a tumor in an accessible location, we will ask for consent from the patient to obtain biopsy before and after the therapy to assess the same molecular markers.

ELIGIBILITY:
Inclusion Criteria:

* One prior chemotherapy treatment: use of single chemotherapy or a regimen containing more than one drug. Regimen must have a platinum agent (cisplatin or carboplatin). Prior biological treatment won't be counted as chemotherapy treatment. Chemoradiation or prior induction or adjuvant chemotherapy +/- chemoradiation will constitute one prior chemotherapy regimen. Patients may not have received Docetaxel. Taxol as part of initial therapy is allowed.
* Documented recurrent/progressive disease by radiographic exam (CT scan, MRI, bone scan or CXR), clinical exam (presence of palpable nodes) or biopsy.
* No signs of clinically active brain metastasis or spinal cord compression. If patient has brain metastasis or cord compression, patient will be eligible if stable without deterioration of performance status after radiation therapy and off corticosteroids.
* Cases with pleural effusion must have another site of disease for measurement and follow-up.
* ECOG performance status 0-1
* Bi-dimensional measurable disease (≥ 1 cm by CT or other radiogram; physical exam alone is permissible if there is no radiographically measurable tumor)
* Laboratory: ANC ≥ 1,500/mm3, Hemoglobin > 8g/dl, platelet ≥ 100,000/mm3, Total Bilirubin ≤ 1.5 mg/dl, Creatinine ≤ 2.0 mg/dl, Transaminase (AST/ALT) ≤ 2.5 X upper normal limit if ALK phosphatase is ≤ Upper normal limit OR ALK may be up to 4X ULN if transaminase are ≤ ULN.
* Age ≥ 18 years old
* Histologic or cytologic diagnosis of NSCLC, biopsy at diagnosis or on recurrence. Histology may include large cell, squamous cell, undifferentiated, bronchioalveolar or adenocarcinoma but not small cell lung cancer or mixed small and non-small cell lung cancer, or carcinoid. Mixed histology non-small cell lung cancer will be allowed, i.e.: large cell neuroendocrine carcinoma.
* IHC of the biopsy specimen, if available, for PDGF-R. Insufficient tissue will not preclude study enrollment.
* FEV1>800 cc

Exclusion Criteria:

* ECOG performance status 2 or worse
* Psychological, familial, sociological or geographical conditions, which prevent weekly medical follow-up or compliance with the study protocol
* Radiation to more than 30% of bone marrow
* More than 1 different prior cytotoxic chemotherapy regimen
* Co-Morbid condition that would affect survival: grade III/IV cardiac problems as defined by New York Heart Association (e.g. end-stage congestive heart failure, myocardial infarction within 6 months of study), random uncontrolled blood sugar ≥300 mg/dl, unstable angina, active infection on antibiotics, FEV1 less than 800 cc, patient with known chronic liver disease (i.e., chronic active hepatitis and cirrhosis)
* Use of investigational agents or chemotherapy within 4 weeks
* Pregnant or nursing women and women or men with reproductive potential unless using effective contraception throughout study and for 3 months after discontinuation of study drug.
* No other active invasive cancer. Patient is < 5 years free of another malignancy except for: other primary malignancy isn't currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Patients with a history of hypersensitivity to taxane, Polysorbate 80 or gemcitabine and who could not tolerate treatment even with 24 H premedication with Decadron and Benadryl. (If the patient had prior hypersensitivity, but did not receive 24 H premedication for taxane, the patient may be eligible if he/she tolerates one cycle with 24 H premedication).
* Existing peripheral neuropathy CTC Version 3> grade 2
* Patient has known diagnosis of human immunodeficiency virus (HIV) infection
* Patients who can not take oral medication. Percutaneous gastrostomy feeding tube will be allowed if Gleevec can be given through PEG
* Patient who had major surgery within 2 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Response rate | Every 2 cycles of therapy and followup

SECONDARY OUTCOMES:
Time to progression, survival and correlation of PDGF and PDGFR with outcome. | Baseline, at completion of therapy, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chao H Huang, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - VA Medical Center, Kansas City, Missouri